CLINICAL TRIAL: NCT01093534
Title: A Study to Evaluate the Overall Effect of Solifenacin 5mg and 10mg on Bladder Wall Thickness and Urinary Nerve Growth Factor in Female Subjects With Overactive Bladder and a Diagnosis of Detrusor Overactivity - A Double-blind, Randomised, Placebo-controlled, Parallel Group, Multi-centre Study.
Brief Title: Study of 2 Doses of Solifenacin Succinate in Female Subjects With Overactive Bladder.
Acronym: SHRINK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 905-EC-007; 2008-005215-17 (EudraCT Number)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Detrusor Overactivity; Overactive Bladder
Keywords: Vesicare; Solifenacin; Detrusor Overactivity; Urinary Nerve Growth Factor; Overactive Bladder; Bladder wall thickness
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received 2 placebo tablets once daily for 12 weeks.
  Interventions: Drug: Placebo
- Solifenacin 5 mg (Experimental): Participants received one 5 mg solifenacin tablet and one placebo tablet, once daily for 12 weeks.
  Interventions: Drug: Placebo; Drug: solifenacin
- Solifenacin 10 mg (Experimental): Participants received two 5 mg solifenacin tablets once daily for 12 weeks.
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: Placebo — Matching solifenacin placebo tablet
  Arms: Placebo; Solifenacin 5 mg
Drug: solifenacin — Tablet for oral administration
  Other Names: YM905; Vesicare
  Arms: Solifenacin 10 mg; Solifenacin 5 mg

SUMMARY:
The purpose is to see if solifenacin has any effect on bladder wall thickness and urine inflammatory marker measurements after 12 weeks of treatment.

DETAILED DESCRIPTION:
Participants satisfying all selection criteria at the end of the 2-week, single blind, placebo run-in period were randomized to receive 12-week double-blind treatment with solifenacin 5 mg or 10 mg once daily, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder (OAB), including urinary frequency, urgency or urge incontinence, for greater than or equal to 3 months
* Urodynamic diagnosis of detrusor overactivity (DO)
* Either naïve to anti-muscarinic treatment (i.e. no prior history of use of anti-muscarinic agents) or 6-months anti-muscarinic treatment free (i.e. have had no anti-muscarinic treatment within 6 months) prior to the screening visit
* Bladder post-void residual volume of less than 30 ml
* Available to complete the study

Exclusion Criteria:

* History of stress urinary incontinence, urethral sphincter incompetence or neurogenic detrusor overactivity
* History, signs or symptoms suggestive of urinary tract infection (confirmed by positive urine analysis), obstruction or urogenital pro-lapse (greater than grade II)
* History of urinary tract operation within 6 months prior to screening
* Indwelling catheter or permanent catheter fitted
* History of pelvic area radiotherapy treatment
* Uncontrolled diabetes mellitus
* History of fibromyalgia
* Post-partum or breast-feeding within 3 months prior to screening visit
* Either pregnant or intends to become pregnant during the study or sexually active, of childbearing potential and is unwilling to utilize a reliable method of birth control (note: reliable methods are contraceptive pills of combination type, hormonal implants or injectable contraceptives)
* Positive pre-study hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus (HIV) result at time of screening
* History of drug and / or alcohol abuse at time of screening
* History of urinary retention, severe gastrointestinal obstruction (including paralytic ileus or intestinal atony or toxic megacolon or severe ulcerative colitis), myasthenia gravis, uncontrolled narrow angle glaucoma or shallow anterior chamber or deemed to be at risk for these conditions
* Undergoing hemodialysis or has severe renal impairment or moderate hepatic impairment or who are on treatment with a potent cytochrome p450 (CYP) 3A4 inhibitor, e.g. Ketoconazole
* Currently dosing with medication(s) intended to treat overactive bladder symptoms or has a history of non-drug treatment, such as electrical therapy, magnetic field stimulation, pelvic floor treatment or bladder training intended to treat overactive bladder symptoms within 6 months prior to screening, as described in the list of prohibited medications
* Currently receiving or has a history of treatment with alpha blockers, botulinum toxin (cosmetic use is acceptable), resiniferatoxin or pelvic floor muscle relaxants within 9 months prior to screening
* Participated in any clinical study less than or equal to 3 months prior to screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2011-06-23 (Actual); Study Completion 2011-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (59):
- United States (2):
  - New York, New York
  - West Reading, Pennsylvania
- Austria (2):
  - Graz
  - Linz
- Belgium (3):
  - Edegem
  - Ghent
  - Kortrijk
- Bulgaria (2):
  - Sofia
  - Varba
- Canada (7):
  - Victoria, British Columbia
  - Barrie, Ontario
  - Brampton, Ontario
  - Brantford, Ontario
  - Kitchener, Ontario
  - Toronto, Ontario
  - Sherbrooke, Quebec
- Czechia (3):
  - Brno
  - Hradec Králové
  - Podolí
- France (2):
  - Marseille
  - Paris
- Germany (4):
  - Aachen
  - Berlin
  - Hanover
  - Munich
- Hungary (3):
  - Budapest
  - Szeged
  - Székesfehérvár
- Israel (3):
  - Haifa
  - Petah Tikva
  - Ramat Gan
- Italy (4):
  - Avellino
  - Milan
  - Rome
  - Varese
- Norway (4):
  - Arendal
  - Drammen
  - Haugesund
  - Tønsberg
- Poland (3):
  - Bydgoszcz
  - Krakow
  - Warsaw
- Timișoara, Romania
- Russia (4):
  - Moscow
  - Nizhny Novgorod
  - Saint Peterburg
  - Yaroslavl
- Slovakia (3):
  - Bardejov
  - Martin
  - Žilina
- Spain (2):
  - Barcelona
  - Madrid
- Sweden (2):
  - Lund
  - Stockholm
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Kocaeli
- United Kingdom (2):
  - Harrow
  - London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg
Started | 186 | 183 | 178
Received Study Treatment | 186 | 182 | 175
Completed | 176 | 167 | 169
Not Completed | 10 | 16 | 9
Not completed — Adverse Event | 2 | 5 | 2
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 7 | 2
Not completed — Other | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all randomized participants who took at least 1 dose of the randomized study medication and for whom any data was reported after the first dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Total
Number analyzed (Participants) | 186 | 182 | 175 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.0) | 55.5 (13.0) | 55.5 (13.3) | 54.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 182 | 175 | 543
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 177 | 177 | 165 | 519
  Black or African American | 1 | 1 | 2 | 4
  Asian | 4 | 1 | 2 | 7
  Other | 4 | 3 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Bladder Wall Thickness
Description: Bladder wall thickness (BWT) measurements were obtained using transvaginal ultrasound. The BWT was derived as one mean value per image pooled over measurements of 3 locations (anterior wall, dome and trigone), and performed by 2 central readers and 1 adjudicator.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT): all randomized participants who received at least 1 dose of randomized study medication and who had a mean BWT measurement at Baseline. Analysis includes participants with available data; Last observation carried forward (LOCF) of post-baseline data was used for imputation of missing values.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Pooled Solifenacin: Participants received either 5 mg or 10 mg solifenacin once daily for 12 weeks.
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 168 | 160 | 150 | 310
mm | 0.00 (1.26) | -0.29 (1.37) | -0.18 (1.18) | -0.24 (1.28)
Statistical Analysis 1: Comparison: Placebo vs Pooled Solifenacin; The null hypothesis was that the mean change from Baseline in BWT in the pooled solifenacin group and placebo was the same. Estimated as two-sided contrast with 95% confidence interval. Power was planned for 80% (assumption: mean difference = 0.5 mm, standard deviation=1.65, 314 and 157 participants, bonferroni adjustment for alpha =0.025); Test type: Superiority or Other; p = 0.095, ANCOVA — Hochberg Method for controlling the overall risk of type I error of 5% was used to adjust for using two co-primary endpoints; ANCOVA model with fixed effects for treatment and region and Baseline of least squares mean BWT as a covariate; Least squares mean difference = -0.169, 95% CI 2-sided [-0.368 to 0.030]

2. Primary Outcome: Neutralized Urinary Nerve Growth Factor Normalized by Urine Creatinine at Week 12
Description: Free (neutralized) urinary nerve growth factor (uNGF) and creatinine (Cr) were measured from urine samples by the central laboratories. Free (neutralized) uNGF/Cr was derived by dividing free (neutralized) uNGF concentrations [pg/mL] by the urine creatinine concentrations (µmol/mL) from the same participant.
Time Frame: Week 12
Population: Full Analysis Set urinary Nerve Growth Factor subset (FAS_uNGF0): all randomized participants who received at least 1 dose of randomized study medication and who had an uNGF/Cr measurement at Baseline and on at least 1 visit thereafter, excluding participants with Baseline uNGF below or equal to the laboratory quantification limit. LOCF was used.
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 176 | 175 | 169 | 344
pg/µmol | 30.359 (26.1760) | 31.855 (29.4371) | 38.917 (60.3231) | 35.325 (47.2694)
Statistical Analysis 1: Comparison: Placebo vs Pooled Solifenacin; The null hypothesis for the co-primary treatment comparison was that the mean free (neutralized) uNGF/Cr value in the pooled solifenacin group and placebo was the same. Wilcoxon rank-sum test was used instead of a contrast from analysis of covariance (ANCOVA), because data was not normally distributed. Power was planned for 80% (assumption: mean difference = 0.74 pg/μmol, standard deviation=2.0, 220 and 110 participants, bonferroni adjustment for alpha =0.025); Test type: Superiority or Other; p = 0.250, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Nonparametric Wilcoxon rank-sum test does not adjust for other factors

3. Secondary Outcome: Total Urinary Nerve Growth Factor Normalized by Urine Creatinine at Week 12
Description: Total (acidified) urinary nerve growth factor (uNGF) and creatinine (Cr) were measured from urine samples by the central laboratories. Total uNGF/Cr was derived by dividing total uNGF concentrations [pg/mL] by the urine creatinine concentrations (µmol/mL) from the same participant.
Time Frame: Week 12
Population: Full Analysis Set urinary Nerve Growth Factor subset (FAS_uNGF0) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 176 | 173 | 169 | 342
pg/µmol | 26.564 (23.0347) | 30.135 (47.4089) | 34.199 (56.2180) | 32.143 (51.9123)

4. Secondary Outcome: Brain Derived Neurotrophic Factor Normalized by Urine Creatinine (uBDNF/Cr) at Week 12
Description: Brain derived neurotrophic factor (uBDNF) and creatinine (Cr) were measured from urine samples by the central laboratories. uBDNF/Cr was derived by dividing uBDNF concentrations [pg/mL] by the urine creatinine concentrations (µmol/mL) from the same participant.
Time Frame: Week 12
Population: Full Analysis Set urinary Brain Derived Neurotrophic Factor (FAS_uBDNF): all randomized participants who received at least 1 dose of randomized study medication, who had given consent for additional analysis and who had an uBDNF/Cr measurement at baseline and on at least 1 visit thereafter. LOCF was used.
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 170 | 170 | 166 | 336
pg/µmol | 116.9 (260.5) | 158.1 (483.0) | 160.4 (373.0) | 159.2 (431.6)

5. Secondary Outcome: Change From Baseline to Week 6 and Week 12 in Bladder Wall Thickness
Description: as for outcome 1
Time Frame: Baseline, Week 6 and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data at each time point (indicated by n).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 155 | 326
mm
  Week 6 (n=157, 145, 141, 286) | -0.01 (1.16) | -0.04 (1.27) | -0.14 (1.15) | -0.09 (1.21)
  Week 12 (n=160, 143, 135, 278) | 0.02 (1.28) | -0.26 (1.37) | -0.22 (1.18) | -0.24 (1.28)

6. Secondary Outcome: Change From Baseline to Week 6 and Week 12 in Neutralized Urinary Nerve Growth Factor Normalized by Urine Creatinine
Description: as for outcome 2
Time Frame: Baseline, Week 6 and Week 12
Population: Full Analysis Set urinary Nerve Growth Factor subset (FAS_uNGF0) participants with available data at each time point (indicated by n).
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 176 | 175 | 169 | 344
pg/µmol
  Week 6 (n=168, 163, 160, 323) | -4.638 (30.7301) | 4.650 (38.3159) | 4.309 (89.1963) | 4.481 (68.3171)
  Week 12 (n=173, 171, 166, 337) | -1.318 (27.9927) | 0.801 (33.3120) | 2.625 (44.0319) | 1.699 (38.9150)

7. Secondary Outcome: Change From Baseline to Week 12 in Mean Number of Events (Micturitions Plus Incontinence Episodes) Per 24 Hours
Description: The average number of micturitions (urinations) and incontinence episodes (any involuntary leakage of urine) per day was derived from the number of events recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 144 | 137 | 122 | 259
events | -1.40 (3.00) | -2.44 (3.55) | -1.80 (2.63) | -2.13 (3.16)

8. Secondary Outcome: Change From Baseline to Week 12 in Mean Number of Urgency Events Per 24 Hours
Description: The intensity of urgency of each micturition (urination) and incontinence episode (any involuntary leakage of urine) was recorded by the participant in an electronic diary according to the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. An urgency event is defined as any micturition or incontinence episode classified by the participant as a grade 3 or 4 on the PPIUS scale. The average number of urgency events per day is derived from the diary data completed by participants on the 3 days prior to the Baseline and Week 12 visits.
Time Frame: 12 weeks
Population: Full analysis set participants with events at Baseline and with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: urgency events
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 139 | 133 | 124 | 257
urgency events | -1.58 (3.04) | -2.22 (3.09) | -1.88 (2.71) | -2.06 (2.91)

9. Secondary Outcome: Change From Baseline to Week 12 in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (urinations) per 24 hours was derived from the number of micturitions recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 144 | 137 | 122 | 259
micturitions | -1.18 (3.03) | -1.80 (3.77) | -1.28 (2.61) | -1.55 (3.28)

10. Secondary Outcome: Change From Baseline to Week 12 in Mean Number of Urgency Micturitions Per 24 Hours
Description: An urgency micturition is defined as any micturition classified by the participant as a grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The average number of urgency micturitions per 24 hours was derived from the number of urgency micturitions recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full Analysis Set participants with urgency micturitions at Baseline and with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: urgency micturitions
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 137 | 130 | 117 | 247
urgency micturitions | -1.35 (2.86) | -1.77 (2.99) | -1.60 (2.45) | -1.69 (2.75)

11. Secondary Outcome: Change From Baseline to Week 12 in Mean Number of Incontinence Episodes Per 24 Hours
Description: The average number of incontinence episodes (any involuntary leakage of urine) per 24 hours was calculated from the number of incontinence episodes recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with incontinence events at Baseline and with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 67 | 62 | 74 | 136
incontinence episodes | -0.60 (1.65) | -1.49 (1.65) | -1.04 (1.76) | -1.24 (1.72)

12. Secondary Outcome: Change From Baseline in Mean Number of Urgency Incontinence Episodes With PPIUS Grade 3 or 4 Per 24 Hours
Description: An urgency incontinence episode is defined as any incontinence episode classified by the participant as a grade 3 or 4 on the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The average number of grade 3 or 4 urgency incontinence episodes per 24 hours was calculated from the number of urgency incontinence episodes recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with grade 3 or 4 urgency incontinence events at Baseline and with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: urgency incontinence episodes
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 59 | 56 | 69 | 125
urgency incontinence episodes | -0.71 (1.52) | -1.32 (1.63) | -0.90 (1.23) | -1.09 (1.43)

13. Secondary Outcome: Change From Baseline in Mean Number of Urgency Incontinence Episodes With PPIUS Grade 4 Per 24 Hours
Description: An urgency incontinence episode is defined as any incontinence episode classified by the participant as a grade 4 on the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The average number of grade 4 urgency incontinence episodes per 24 hours was calculated from the number of urgency incontinence episodes recorded by the participant in an electronic diary for 3 days before the Baseline and Week 12 clinic visits.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with grade 4 urgency incontinence events at Baseline and with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: urgency incontinence episodes
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 50 | 49 | 61 | 110
urgency incontinence episodes | -0.70 (1.46) | -0.96 (0.91) | -0.70 (1.16) | -0.82 (1.06)

14. Secondary Outcome: Change From Baseline to Week 12 in Mean Level of Urgency
Description: The intensity of urgency of each micturition (urination) and incontinence episode (any involuntary leakage of urine) was recorded by the participant in an electronic diary according to the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The mean level of urgency was calculated by adding the PPIUS grade for all events (micturition or incontinence) and dividing by the number of episodes recorded in the diary over 3 days prior to the Baseline and Week 12 visits.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 144 | 137 | 122 | 259
units on a scale | -0.15 (0.525) | -0.23 (0.504) | -0.24 (0.578) | -0.23 (0.539)

15. Secondary Outcome: Change From Baseline to Week 12 in Total Urgency Score
Description: The intensity of urgency of each micturition (urination) and incontinence episode (any involuntary leakage of urine) was recorded by the participant in an electronic diary according to the Patient Perception of Intensity of Urgency Scale (PPIUS) as follows: 0 = No urgency; 1 = Mild urgency; 2 = Moderate urgency, could postpone voiding a short while; 3 = Severe urgency, could not postpone voiding; 4 = Urge incontinence, leaked before arriving to the toilet. The total urgency score was calculated by adding all PPIUS scores over a 3-day period prior to the Baseline and Week 12 visits for each participant.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 144 | 137 | 122 | 259
units on a scale | -13.61 (25.98) | -22.39 (29.80) | -16.91 (22.57) | -19.81 (26.73)

16. Secondary Outcome: Change From Baseline in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. A negative change from Baseline score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale | -0.7 (1.33) | -1.3 (1.38) | -1.3 (1.26) | -1.3 (1.33)

17. Secondary Outcome: Change From Baseline in Patient Assessment of Urgency Bother
Description: The participants' perception and impression of bother associated with their condition were assessed using the Urgency Bother-Visual Analog Scale (UB-VAS). The participant was asked to place a vertical mark on a 100 mm line to indicate how much bother has urgency been for them in the past week, whereby 'no bother at all' is represented on the left end (score = 0) and 'worst possible bother' (score = 100) at the right end of the line. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale | -12.60 (29.51) | -27.70 (30.39) | -28.90 (28.72) | -28.20 (29.57)

18. Secondary Outcome: Change From Baseline in Patient Assessment of Treatment Satisfaction
Description: The treatment satisfaction visual analog scale (TS_VAS) asks patients to rate their satisfaction with treatment by placing a vertical mark on a 100 mm line where the endpoints are labeled 'No, not at all' on the left (score = 0) to 'Yes, completely satisfied' on the right (score = 100). A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale | 18.90 (42.18) | 24.90 (39.58) | 31.90 (41.02) | 28.20 (40.36)

19. Secondary Outcome: Percentage of Participants With Improvement and Worsening on the 5 Dimensions of the EQ-5D
Description: The participants' quality of life was assessed using the EuroQoL 5 Dimension Questionnaire (EQ-5D). The EQ-5D is a standardized instrument for use as a measure of health outcome and is based on the following 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. For each dimension participants were asked to select the statement which best described their health that day, from level 1 (indicating no problems) to 3 (indicating extreme problems/unable to perform). Improvement was defined as a change from a state of being unable to perform or extreme problems at Baseline to no problems or to some or moderate problems at Week 12, and from some or moderate problems to no problems. Worsening was defined as a change from no problems at Baseline to some or moderate problems or to a state of being unable to perform or extreme problems at Week 12, and from some or moderate problems to a state of being unable to perform or extreme problems.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 165 | 155 | 146 | 301
percentage of participants
  Mobility: Improvement | 6.7 | 10.3 | 9.6 | 10.0
  Mobility: Worsening | 10.3 | 7.1 | 3.4 | 5.3
  Self-care: Improvement | 2.4 | 3.9 | 3.4 | 3.7
  Self-care: Worsening | 2.4 | 3.2 | 4.1 | 3.7
  Usual Activities: Improvement | 7.9 | 7.7 | 11.0 | 9.3
  Usual Activities: Worsening | 7.9 | 11.0 | 4.8 | 8.0
  Pain/Discomfort: Improvement | 15.2 | 19.4 | 18.5 | 18.9
  Pain/Discomfort: Worsening | 10.3 | 11.0 | 4.8 | 8.0
  Anxiety/Depression: Improvement | 17.0 | 17.4 | 19.9 | 18.6
  Anxiety/Depression: Worsening | 10.3 | 11.0 | 13.7 | 12.3

20. Secondary Outcome: Change From Baseline in EuroQoL 5-Dimension Questionnaire Visual Analog Scale
Description: The participants' quality of life was assessed using the EuroQoL 5 Dimension Questionnaire (EQ-5D) visual analog scale (VAS). Health status is completed by the participant indicating their own health state today by drawing a line on a vertical scale from 0 to 100 where the endpoints are labeled 'Worst imaginable health state' (=0) and 'Best imaginable health state' (=100). On the EQ-5D VAS, a positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale | 3.60 (16.86) | 4.80 (20.22) | 5.10 (17.86) | 4.90 (19.12)

21. Secondary Outcome: Change From Baseline in Symptom Bother Score
Description: Overactive bladder symptoms were assessed using the symptom bother scale of the Overactive Bladder Symptom and Health-Related Quality of Life Questionnaire (OAB-q). The OAB-q is a patient-administered instrument comprising an 8-item symptom bother scale and 25 health-related quality of life items (see next outcome measure). In the symptom bother scale participants were asked how much they had been bothered by selected bladder symptoms during the past 4 weeks. Each question has a 6-point Likert scale response ranging from 'not at all' (1) to 'a very great deal' (6). The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from Baseline in symptom bother score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale | -14.90 (19.11) | -22.32 (20.59) | -22.91 (18.69) | -22.60 (19.69)

22. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQL)
Description: Health-related quality of life was assessed by the Overactive Bladder Symptom and Health-Related Quality of Life Questionnaire (OAB-q). The OAB-q is a patient-administered instrument comprising of an 8-item symptom bother scale (see previous outcome measure) and 25 HRQL items comprising 4 subscales (concern, coping, social interaction and sleep) and a total HRQL score. Participants were asked how their overall bladder symptoms had affected their life in the past 4 weeks. Each of the 25 HRQL questions has a 6-point Likert scale response ranging from 'none of the time' (1) to 'all of the time' (6). The HRQL subscale scores were calculated by summing the responses of the items within each subscale.The HRQL total score was calculated by adding the 4 HRQL subscale scores,. All scores were transformed to a scale from 0 to 100 where higher scores indicate better quality of life. A positive change from Baseline in HRQL score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
units on a scale
  Total score | 11.72 (16.71) | 17.25 (19.74) | 17.69 (15.75) | 17.46 (17.94)
  Coping subscale | 12.40 (18.85) | 18.26 (20.89) | 20.21 (19.42) | 19.18 (20.20)
  Concern subscale | 13.80 (18.64) | 20.35 (22.52) | 20.77 (18.73) | 20.55 (20.79)
  Sleep subscale | 10.80 (19.31) | 15.50 (21.33) | 15.10 (15.95) | 15.30 (18.95)
  Social interaction subscale | 8.70 (16.95) | 13.00 (19.65) | 12.00 (15.54) | 12.50 (17.81)

23. Secondary Outcome: Change From Baseline to Week 12 in Brain Derived Neurotrophic Factor Normalized by Urine Creatinine (uBDNF/Cr)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: Full Analysis Set urinary Brain Derived Neurotrophic Factor (FAS_uBDNF); LOCF was used.
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 170 | 170 | 166 | 336
pg/µmol | -27.4 (317.6) | 31.1 (426.9) | -88.1 (980.6) | -27.8 (754.4)

24. Secondary Outcome: Change From Baseline to Week 12 in Total Urinary Nerve Growth Factor Normalized by Urine Creatinine
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: Full Analysis Set urinary Nerve Growth Factor subset (FAS_uNGF0) participants with available data; LOCF was used.
Measure: Mean (Standard Deviation); unit: pg/µmol
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 176 | 173 | 169 | 342
pg/µmol | -0.962 (24.2241) | 2.758 (49.0191) | 3.858 (44.0421) | 3.302 (46.5612)

25. Secondary Outcome: Percentage of Participants With Improvement or Deterioration in Patient Perception of Bladder Condition (PPBC)
Description: The PPBC scale is a global assessment tool that asks patients to rate their impression of their current bladder condition on a 6-point scale from 1: 'Does not cause me any problems at all'; 2: 'Causes me some very minor problems'; 3: 'Causes me some minor problems'; 4: 'Causes me (some) moderate problems'; 5: 'Causes me severe problems' and 6: 'Causes me many severe problems'. Improvement: ≥ 1 point improvement compared to Baseline; Major Improvement: ≥ 2 point improvement compared to Baseline; Deterioration: ≥ 1 point deterioration compared to Baseline.
Time Frame: Baseline and Week 12
Population: Full Analysis Set Bladder Wall Thickness (FAS_BWT) participants with available data; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg | Pooled Solifenacin
Number analyzed (Participants) | 175 | 171 | 153 | 324
percentage of participants
  Deterioration | 15.4 | 6.4 | 5.2 | 5.9
  No change | 34.9 | 21.6 | 20.3 | 21.0
  Improvement | 49.7 | 71.9 | 74.5 | 73.1
  Major Improvement | 27.4 | 39.8 | 44.4 | 42.0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Solifenacin 5 mg | Solifenacin 10 mg
Serious Adverse Events (participants affected / at risk) | 1/186 | 1/182 | 4/175
Other Adverse Events (participants affected / at risk) | 9/186 | 21/182 | 34/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Solifenacin 5 mg (N=182) | Solifenacin 10 mg (N=175)
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Endotoxic shock (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Solifenacin 5 mg (N=182) | Solifenacin 10 mg (N=175)
Dry mouth (Gastrointestinal disorders) | 2 | 16 | 30
Constipation (Gastrointestinal disorders) | 7 | 8 | 9

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the currency or completeness of the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 60 days prior to publication for review and comment. Sponsor may delay the publication for up to 6 months to seek patent protection.